CLINICAL TRIAL: NCT00713011
Title: Randomized Open-label 2-arm Parallel Design Comparator Study of the Effect of Adalat® XL® Compared to Diltiazem on Proteinuria and Blood Pressure in Patients With Diabetes and Mild to Moderate Hypertension When Used as an Add on to Avalide®
Brief Title: Adalat XL vs Diltiazem on Proteinuria and Blood Pressure in Hypertensive Diabetic Patients
Acronym: CARDINAL
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was stopped by sponsor prior to first patient assignment to groups due to operational reasons.
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Healthcare Pharmaceuticals Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12716
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Diabetic Nephropathies; Hypertension
Keywords: Adalat XL; Diltiazem; Tiazac XC; Proteinuria
MeSH Terms: conditions — Diabetic Nephropathies; Hypertension; Proteinuria | interventions — Nifedipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Adalat XL
- Arm 2 (Active Comparator)
  Interventions: Drug: Tiazac XC

INTERVENTIONS:
Drug: Adalat XL — Patients will receive Avalide (Irbesartan/ hydrochlorothiazide; 300 mg/12.5 mg per day or 300 mg/25.0 mg per day) during the 12 week screening period and during the 18 week treatment period. At baseline, patients will be provided with Adalat XL at a starting dose of 20 or 30 mg. Adalat XL will be titrated during the 18 week treatment period in order to optimize blood pressure. Adalat XL will be supplied in 20 mg, 30 mg, 60 mg, and 90 mg.
  Arms: Arm 1
Drug: Tiazac XC — Patients will receive Avalide (Irbesartan/ hydrochlorothiazide; 300 mg/12.5 mg per day or 300 mg/25.0 mg per day) during the 12 week screening period and during the 18 week treatment period. At baseline, patients will be provided with Tiazac XC at a starting dose of 180 mg. Tiazac XC will be titrated during the 18 week treatment period in order to optimize blood pressure. Tiazac XC will be supplied in 180 mg, 240 mg, 300 mg and 360 mg.
  Arms: Arm 2

SUMMARY:
The study consists of a 12 week run-in period when all subjects are stabilized on a single dose of Avalide (300 mg/12.5 mg or 300mg/25mg dose) per day. After this 12 week run-in ends, subjects will be randomly assigned to start the addition of either Adalat XL or Tiazac XC for 18 weeks of treatment. Subjects will have a 1 in 2 chance of receiving the study drug Adalat XL and a 1 in 2 chance of receiving the drug Tiazac XC. An end of treatment visit will be done 18 weeks after start of study drug. The expected duration of the study is 30 weeks. The purpose of this study is to compare the change in proteinuria, through a urine test, while taking study drug until high blood pressure (BP) is reduced to near normal levels in study subjects with diabetic nephropathy and hypertension.

ELIGIBILITY:
Inclusion Criteria:

* >/= 18 and < 80 years old.
* Diagnosed with hypertension.
* Diagnosed with diabetes mellitus type 2 for at least 6 mths prior to entry and on stable medication for diabetes for at 1 mth prior to screening.
* Treated on ARB, ACE inhibitor with or without hydrochlorothiazide and suitable to receive combination therapy with Avalide at 300mg/12.5mg per day or 300mg/25mg per day.
* Diagnosed with diabetic nephropathy and have proteinuria between 0.8g/day and 5.0g/day at screening and then between 0.8g/day and 3.0g/day at randomization.
* Medically appropriate to receive Adalat XL or Tiazac XC.

Exclusion Criteria:

* History of alcohol or substance abuse.
* Significant CV disorder such as ischemic heart disease, arrhythmias within the last 6 mths, or any history of severe congestive heart failure.
* Myocarditis or pericarditis within last 30 day of screening.
* ECG showing evidence of major arrhythmia or conduction disturbances requiring treatment with anti-arrhythmic medication.
* Females with child-bearing potential or males with a partner of child-bearing potential unless willing to use effective contraception during the study and 3 mths after the end of study.
* Females who are pregnant, lactating or planning pregnancy during the study and for 3 mths after the study end.
* Known hypersensitivity to Adalat XL or Tiazac XC or other calcium channel blockers of the dihydropyridine class.
* Resting heart rate <50 or >110 bpm.
* Presence of secondary or malignant hypertension.
* DBP >/= 180 and/or SBP >/= 110 mmHg.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2009-03 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Change in Proteinuria | Baseline/Randomization to Week 18

SECONDARY OUTCOMES:
Percentage of subjects reaching a BP target of 130/80 mmHg at Week 18 | Baseline/Randomization to Week 18
Number and doses of anti-hypertensives used in the 2 treatment arms | Baseline/Randomization to Week 18
Levels of urinary albumin and protein content and estimated glomerular filtration rate (GFR) in the 2 treatment groups | Baseline/Randomization to Week 18
Early BP reduction from randomization achieved with the starting dose in the 2 treatment arms | Baseline/Randomization to Week 1
Adverse Events leading to early withdrawal | Screening to end of study
All Adverse Events especially, edema | Screening to end of study
Change in index of glycemia (HbA1c) | Screening to Week 18

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer